CLINICAL TRIAL: NCT07307781
Title: Clinical and dEmographic chaRacteristics of Patients With Frequent COPD Exacerbations and Evaluation of Therapeutic Approaches in Treatment in Moscow
Brief Title: Study of Patient With Frequent Exacerbations in Moscow
Acronym: CERERA-MOSCOW
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00217
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Study is multicenter, non-interventional, ambispective registry to evaluate the demographic and clinical characteristics, therapeutic approaches and outcomes in COPD outpatients with frequent exacerbations in Moscow

DETAILED DESCRIPTION:
This ambispective study consists of retrospective and prospective parts:

* Retrospective part aims to describe the demographic and clinical characteristics, as well as therapeutic approaches in COPD outpatients with frequent exacerbations during the 52 weeks prior to screening;
* Prospective part aims to evaluate current therapeutic approaches for such patients and their outcomes in real-world clinical practice.

The patient participation in the study will include two visits:

* Visit 1 - baseline: inclusion into the study, retrospective collection of medical history and data on COPD course and treatment during the previous 52 weeks, and primary data collection trough patient interview and physician assessment;
* Visit 2 - follow-up at Week 24 (±6): primary data collection trough patient interview and physician assessment.

All visits will be conducted by a study physician in accordance with routine clinical practice for the observation and management of COPD patients. For each eligible patient, the study physician will collect data in an individual electronic Case Report Form (eCRF) based on source medical documentation.

Expected duration of the inclusion period is 12 months OR until 500 eligible patients are included into the study, whichever occurs first. Overall expected duration of the study (from the first patient inclusion to the last patient last visit) is approximately 25 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of inclusion;
2. Signed and dated written informed consent in accordance with ICH GCP and local law prior to inclusion in the study;
3. Confirmed diagnosis of moderate-to-very severe (GOLD 2-4) COPD established by spirometry demonstrating a post-bronchodilator ratio of forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) <0.7 obtained outside an exacerbation;
4. ≥2 moderate or ≥1 severe COPD exacerbations in previous 52 weeks;
5. Dual inhaled maintenance therapy (LABA/LAMA, ICS/LAMA, or ICS/LABA) for at least 6 weeks prior to screening

Exclusion Criteria:

1. Current or previous treatment with triple combination (ICS/LAMA/LABA) as maintenance therapy within 52 weeks prior to screening visit;
2. COPD due to documented alpha-1-antitrypsin deficiency;
3. A diagnosis of bronchiectasis, sarcoidosis, interstitial lung diseases, or idiopathic pulmonary fibrosis, exacerbation of asthma or any acute or chronic disease that, as deemed by Investigator, limits the ability of patients to participate in this study or could influence the interpretation of the results;
4. The participation in any interventional clinical study currently or within 52 weeks prior to inclusion; participation in non-interventional, observational registries without protocol-driven treatment changes does not constitute an exclusion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study population consists of 500 adult patients with moderate-to-very severe COPD who have experienced ≥2 moderate or ≥1 severe exacerbations within the previous 52 weeks and received dual inhaled maintenance therapy (LABA/LAMA, ICS/LAMA, or ICS/LABA combinations, but not triple ICS/LAMA/LABA therapy) for at least 6 weeks prior to screening
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
To describe the baseline mean age of outpatients with COPD in Moscow. | 52 weeks of retrospective data before visit 1
  1. Mean age (years) at inclusion, and proportion of patients within different age groups:
     1. <50 years;
     2. 50-65 years;
     3. >65 years;
  2. Mean age (years) at the primary COPD diagnosis;
To describe the baseline Demographic data characterisics of outpatients with COPD in Moscow. | 52 weeks of retrospective data before visit 1
  3. Proportion of men and women; 4. Proportion of patients with different educational status at inclusion:
  1. Higher education;
  2. Secondary special education;
  3. Secondary general education.
To describe the baseline Negative lifestyle factors of outpatients with COPD in Moscow. | 52 weeks of retrospective data before visit 1
  5. Proportion of patients with different negative lifestyle factors at inclusion (evaluated at Visit 1 based on patient interview):
  a. Proportion of patients with history of smoking (former smokers) and current smokers - applicable for both tobacco and e-cigarettes (vapes) smokers; d. Proportion of patient with physical inactivity. 7. Proportion of overweight patients
To describe the baseline Anthropometry data characterisics of outpatients with COPD in Moscow. | 52 weeks of retrospective data before visit 1
  6. Mean body mass index (BMI) (kg/m2) at inclusion (evaluated at Visit 1 or the most recent available value obtained within the previous 52 weeks if cannot be measured at Visit 1);
To describe the baseline mean smoking index . | 52 weeks of retrospective data before visit 1
  5 b. applicable for former and current tobacco smokers;
To describe the baseline mean duration of smoking | 52 weeks of retrospective data before visit 1
  5 c. applicable for former and current e cigarettes (vapes) smokers;
To describe a COPD clinical course of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  8. Proportion of patients with different COPD severity based on GOLD classification at inclusion:
  1. GOLD 2 (moderate);
  2. GOLD 3 (severe);
  3. GOLD 4 (very severe); 9. Proportion of patients who have experienced at least 1 moderate COPD exacerbation during 52 weeks prior to inclusion; 11. Proportion of patients who have experienced at least 1 severe COPD exacerbation during 52 weeks prior to inclusion; 12. Proportion of patients who have experienced different numbers of severe COPD exacerbations during 52 weeks prior to inclusion:
  a. 0 severe COPD exacerbations; b. 1 severe COPD exacerbation; c. 2 severe COPD exacerbations; d. ≥3 severe COPD exacerbations;
To describe a COPD exacerbation of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  10. Annualized rate of moderate COPD exacerbations prior to inclusion 13. Annualized rate of severe COPD exacerbations prior to inclusion
To describe a severe COPD exacerbation of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  14. Cumulative days of severe COPD exacerbations prior to inclusion
To describe a COPD drug therapy of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  15. Proportion of patients receiving different classes of drugs for treatment of COPD (both maintenance therapy and exacerbation management) and their combinations (administered either as separate agents or as fixed combination) prior to inclusion:
  1. Short-Acting β2-Adrenergic Agonist (SABA) alone;
  2. ICS alone;
  3. LABA alone;
  4. LAMA alone;
  5. LABA/LAMA;
  6. ICS/LABA;
  7. ICS/LAMA;
  8. LABA/LAMA plus:
  a) Macrolide antibiotics; b) Systemic corticosteroids.
To describe a Spirometry parameters at baseline of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  16. Mean pre-bronchodilator FEV1 at inclusion (the most recent available value obtained within the previous 52 weeks outside of an exacerbation); 17. Mean post-bronchodilator FEV1 at inclusion (the most recent available value obtained within the previous 52 weeks outside of an exacerbation); 18. Mean FVC at inclusion (the most recent available value obtained within the previous 52 weeks outside of an exacerbation);
To describe a FEV1 / FVC ratio at baseline of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  19. Mean post-bronchodilator FEV1 / FVC ratio at inclusion (the most recent available value obtained within the previous 52 weeks outside of an exacerbation).
To describe Blood eosinophils count at baseline of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  20. Mean blood eosinophils count (cells/μl) at inclusion (the most recent available value obtained within the previous 52 weeks); 21. Proportion of patients with different levels of blood eosinophils count at inclusion (based on the most recent available value obtained within the previous 52 weeks):
  1. <150 cells/μl;
  2. 150-300 cells/μl;
  3. ≥301 cells/μl.
To describe CAT questionnaire score at baseline of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  22. Mean COPD Assessment Test (CAT) score at inclusion (evaluated at Visit 1 or the most recent available value obtained within the previous 6 weeks if evaluation at Visit 1 is not possible).
To describe Healthcare resource utilization of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  23. Proportion of patients with healthcare resource utilization events during 52 weeks prior to inclusion:
  1. Unscheduled outpatient visits due to COPD;
  2. Emergency department visits / emergency calls due to COPD;
  3. Hospitalizations:
  a) Any hospitalizations; b) COPD-related hospitalizations; c) Hospitalizations due to respiratory reason; d) Hospitalizations due to cardiovascular reason; e) Hospitalizations due to other reason; 24. Mean duration of COPD-related hospitalizations (days) during 52 weeks prior to inclusion; 25. Proportion of patients with COPD-related disability at inclusion:
  1. Any disability;
  2. I disability group;
  3. II disability group;
  4. III disability group
To describe COPD comorbidities at baseline of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  26. Proportion of patients with different comorbidities at inclusion (diagnosed by study physician at Visit 1 or diagnosed at any time previously and recorded based on medical documentation or patient interview):
  1. Heart failure
  2. Ischemic heart disease
  3. Myocardial infarction
  4. Arrhythmia
  5. Stroke
  6. Arterial hypertension
  7. Peripheral arterial disease
  8. Diabetes mellitus (type I, type II)
  9. Chronic kidney disease
  10. Pulmonary hypertension
  11. Pulmonary embolism
  12. Another comorbidity 27. Proportion of patients with different types of arrythmia at inclusion (to be calculated in the subgroup of patients with any arrhythmia before or at Visit 1):
  a. Atrial fibrillation / atrial flutter; b. Ventricular arrhythmia; c. Another arrhythmia;
To describe COPD and Heart Failure comorbidity at baseline of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  28. Proportion of patients with each HF phenotype based on left ventricle ejection fraction (LVEF) at inclusion (to be calculated in the subgroup of patients with any HF before or at Visit 1):
  1. HF with reduced ejection fraction (HFrEF);
  2. HF with mid-range ejection fraction (HFmrEF);
  3. HF with preserved ejection fraction (HFpEF);
To describe LVEF at baseline of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  29. Mean and median LVEF (%) at inclusion (to be calculated in the subgroup of patients with any HF before or at Visit 1 and available data on LVEF based on echocardiography);
To describe COPD and Chronic Kidney Disease comorbidity at baseline of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  30. Proportion of patients with each CKD stage based on estimated glomerular filtration rate (eGFR) at inclusion (to be calculated in the subgroup of patients with any CKD before or at Visit 1):
  1. Stage C1 (eGFR ≥90 ml/min/1.73 m2);
  2. Stage C2 (eGFR 89-60 ml/min/1.73 m2);
  3. Stage C3a (eGFR 59-45 ml/min/1.73 m2);
  4. Stage C3b (eGFR 44-30 ml/min/1.73 m2);
  5. Stage C4 (eGFR 29-15 ml/min/1.73 m2);
  6. Stage C5 (eGFR <15 ml/min/1.73 m2);
To describe COPD and Arterial Hypertension (AH) comorbidity at baseline of outpatients with COPD in Moscow | 52 weeks of retrospective data before visit 1
  31. Proportion of patients with each AH degree at inclusion (to be evaluated in patients with AH diagnosed before or at Visit 1):
  1. 1st degree of AH;
  2. 2nd degree of AH;
  3. 3rd degree of AH; 32. Proportion of patients with each AH stage at inclusion (to be evaluated in patients with AH diagnosed before or at Visit 1):
  a. Stage I; b. Stage II; c. Stage III; 33. Proportion of patients with risk category at inclusion (to be evaluated in patients with AH diagnosed before or at Visit 1):
  1. Low risk;
  2. Intermediate risk;
  3. High risk;
  4. Very high risk;
To describe blood pressure at baseline of outpatients with COPD in Moscow | at visit 1
  34. Mean office systolic blood pressure (SBP) (mmHg) measured at inclusion (in total population and by presence of AH diagnosed before or at Visit 1); 35. Mean office diastolic blood pressure (DBP) (mmHg) measured at inclusion (in total population and by presence of AH diagnosed before or at Visit 1);
To describe a treatment of comorbidities at baseline of outpatients with COPD in Moscow | at visit 1
  36. Proportion of patients receiving different classes of medications used for treatment of comorbidities (to be evaluated in the subgroup of patients with at least one comorbidity specified above in paragraph #26)

SECONDARY OUTCOMES:
To describe COPD drug therapy during the follow-up period and its change compared to the previous 52 weeks | 24 weeks after visit 1
  1. Proportion of patients receiving different classes of drugs for maintenance therapy of COPD and their combinations (administered either as separate agents or as fixed combination) after Visit 1 and at Visit 2:
     1. SABA alone
     2. ICS alone
     3. LABA alone
     4. LAMA alone
     5. LABA/LAMA;
     6. ICS/LABA
     7. ICS/LAMA
     8. LABA/LAMA/ICS
     <!-- -->
     1. Any combination
     2. Open combination
     3. Fixed combination i. Macrolide antibiotics j. Systemic CS:
     <!-- -->
     1. Any regimen
     2. Intermittent regimen
     3. Regular regimen
To describe corticosteroid therapy during the follow-up period of outpatients with COPD in Moscow | 24 weeks after visit 1
  3. Mean systemic CS daily dose (mg/day in prednisolone equivalent) during follow-up period (to be evaluated in the subgroup of patients who have been receiving systemic CS during follow-up period);
To describe changes of inhaled COPD therapy during the follow-up period of outpatients with COPD in Moscow | 24 weeks after visit 1
  4. Proportion of patients with different types of change of inhaled COPD therapy during the follow-up period compared to the 52 weeks prior to inclusion:
  a. Dosage adjustment:
  1. Increase in the dose of one or both components;
  2. Reduction in the dose of one or both components; b. Switch within the same drug class c. Switch between drug classes (dual-to-dual) d. Therapy escalation to triple combination; e. Therapy de-escalation to monotherapy
To describe COPD therapy during the follow-up period of outpatients with COPD in Moscow | 24 weeks after visit 1
  4. Proportion of patients with different types of change of inhaled COPD therapy during the follow-up period compared to the 52 weeks prior to inclusion:
  a. Dosage adjustment:
  1. Increase in the dose of one or both components;
  2. Reduction in the dose of one or both components; b. Switch within the same drug class c. Switch between drug classes (dual-to-dual) d. Therapy escalation to triple combination; e. Therapy de-escalation to monotherapy 5. Proportion of patients who have been receiving systemic CS for COPD exacerbation treatment during the follow-up period
To describe COPD clinical course during the follow-up period and its change compared to the previous 52 weeks of outpatients with COPD in Moscow | 24 weeks after visit 1
  6. Proportion of patients with different COPD severity based on GOLD classification at Visit 2 7. Proportion of patients with COPD progression to more severe GOLD category over the follow-up period 8. Proportion of patients with COPD improvement to less severe GOLD category over the follow-up period overall and by GOLD category at baseline 9. Proportion of patients who have experienced at least 1 COPD exacerbation during the follow-up period; 10. Proportion of patients who have experienced at least 1 moderate COPD exacerbation during the follow-up period 11. Proportion of patients who have experienced at least 1 severe COPD exacerbation during the follow-up period; 12. Proportion of patients who have experienced different numbers of severe COPD exacerbations during the follow-up period
To describe exacerbations of outpatients with COPD in Moscow | 24 weeks after visit 1
  11. Annualized rate of moderate COPD exacerbations during the follow-up period 14. Annualized rate of severe COPD exacerbations during the follow-up period; 15. Cumulative days of severe COPD exacerbations during the follow-up period
To describe Spirometry parameters during follow-up period and their change compared to the previous 52 weeksof outpatients with COPD in Moscow | 24 weeks after visit 1
  16. Mean pre-bronchodilator FEV1 at Visit 2 (the most recent available value obtained within the follow-up period outside of an exacerbation); 17. Mean change of pre-bronchodilator FEV1 from baseline to the end of the follow-up period; 18. Mean post-bronchodilator FEV1 at Visit 2 (the most recent available value obtained within the follow-up period outside of an exacerbation); 19. Mean change of post-bronchodilator FEV1 from baseline to the end of the follow-up period; 20. Mean FVC at Visit 2 (the most recent available value obtained within the follow-up period outside of an exacerbation); 21. Mean change of FVC from baseline to the end of the follow-up period;
To describe Spirometry FEV1 / FVC ratio during follow-up period and their change compared to the previous 52 weeks of outpatients with COPD in Moscow | 24 weeks after visit 1
  22. Mean post-bronchodilator FEV1 / FVC ratio at Visit 2 (the most recent available value obtained within the follow-up period outside of an exacerbation); 23. Mean change of FEV1 / FVC ratio from baseline to the end of the follow-up period
To describe Blood eosinophils count during follow-up period and its change compared to the previous 52 weeks of outpatients with COPD in Moscow | 24 weeks after visit 1
  24. Mean blood eosinophils count (cells/μl) at Visit 2 (the most recent available value obtained within the follow-up period); 25. Mean change in blood eosinophils count (cells/μl) from baseline to the end of the follow-up period;
To describe Proportion of patients with different levels of blood eosinophils count of outpatients with COPD in Moscow | 24 weeks after visit 1
  26. to evaluated at Visit 2 (based on the most recent available value obtained within the follow-up period):
  1. <150 cells/μl;
  2. 150-300 cells/μl;
  3. ≥301 cells/μl.
To describe CAT questionnaire score during follow-up period and its change compared to the previous 52 weeks of outpatients with COPD in Moscow | 24 weeks after visit 1
  27. Mean CAT score at Visit 2 (evaluated at Visit 2 or the most recent available value obtained within the 6-week period prior to Visit 2 if evaluation at Visit 2 is not possible); 28. Mean change of CAT score from baseline to the end of the follow-up period
To describe Proportion of responders based on CAT score of outpatients with COPD in Moscow | 24 weeks after visit 1
  29. defined as proportion of patients who achieved minimal clinically important difference (MCID) of 2 or more points from baseline to the end of the follow-up period.
To describe Healthcare resource utilization during follow-up period and its change compared to the previous 52 weeks of outpatients with COPD in Moscow | 24 weeks after visit 1
  30. Proportion of patients with healthcare resource utilization events during the follow-up period 32. Proportion of patients with COPD-related disability at Visit 2 33. Proportion of patients with newly established COPD-related disability during the follow-up period (to be evaluated in the subgroup of patients with disability absent at inclusion) 34. Proportion of patients with the change of COPD-related disability level during the follow-up period (to be evaluated in the subgroup of patients with disability present at inclusion)
To describe hospitalization during follow-up period and its change compared to the previous 52 weeks of outpatients with COPD in Moscow | 24 weeks after visit 1
  31. Mean duration of COPD-related hospitalizations (days) during the follow-up period
To describe COPD comorbidities during the follow-up period and their change compared to the previous 52 weeks of outpatients with COPD in Moscow | 24 weeks after visit 1
  35. Proportion of patients with newly diagnosed comorbidities at Visit 2 36. Proportion of patients with different types of arrythmia newly diagnosed during the follow-up period 37. Proportion of patients with each HF phenotype based on LVEF newly diagnosed during the follow-up period 39. Proportion of patients with decompensation of previously diagnosed HF 40. Proportion of patients with each CKD stage based on eGFR newly diagnosed during the follow-up period 41. Proportion of patients with each AH degree at Visit 2 42. Proportion of patients with each AH stage at Visit 2 43. Proportion of patients with risk category at Visit 2 46. Proportion of patients receiving different classes of medications used for treatment of comorbidities
To describe disability during follow-up period of outpatients with COPD in Moscow | 24 weeks after visit 1
  32. Proportion of patients with COPD-related disability at Visit 2 33. Proportion of patients with newly established COPD-related disability during the follow-up period (to be evaluated in the subgroup of patients with disability absent at inclusion) 34. Proportion of patients with the change of COPD-related disability level during the follow-up period (to be evaluated in the subgroup of patients with disability present at inclusion)
To describe LVEF during follow-up period of outpatients with COPD in Moscow | 24 weeks after visit 1
  38. Mean and median LVEF (%) (to be calculated in the subgroup of patients with any HF newly diagnosed during the follow-up period and available data on LVEF based on echocardiography);
To describe blood pressure during follow-up period of outpatients with COPD in Moscow | 24 weeks after visit 1
  44. Mean office SBP (mmHg) measured at Visit 2 (in total population and by presence of AH diagnosed at any time); 45. Mean office DBP (mmHg) measured at Visit 2 (in total population and by presence of AH diagnosed at any time);
To describe adverse drug reactions during follow-up period of outpatients with COPD in Moscow | 24 weeks after visit 1
  47. Proportion of patients with adverse drug reactions (ADR) related to COPD treatment during the follow-up period overall and by system organ class (SOC) and preferred term (PT) of Medical Dictionary for Regulatory Activities (MedDRA), by related drug class, by seriousness, by severity and by actions taken regarding ADR and regarding related drug; 48. Proportion of patients who discontinued any COPD treatment due to ADR overall and by drug class discontinued.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Moscow, Russia